CLINICAL TRIAL: NCT03345641
Title: Emotional Reactions of Mothers Facing Premature Births
Acronym: mother's traum
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PR06002
Record Dates: First submitted 2017-10-23; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Premature Birth; Mother's Post-traumatic Reaction; Mother-infant Interactions
Keywords: premature birth; mother's post-traumatic reaction; mother-infant interactions
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- dyads: dyads with babies and their mothers
  Interventions: Other: describe precocious maternal impressions when confronting the premature birth of her infant

INTERVENTIONS:
Other: describe precocious maternal impressions when confronting the premature birth of her infant

SUMMARY:
Our intervention in the maternity and neonatal wards helped our sensibility to the immediate parental reaction to the premature birth. Among these reactions, what is called "stress" by the parents occurs most often and is at the origin of trauma. The investigators can cite the unexpected confrontation with a baby is far from corresponding to what the parents had anticipated; the stunned feeling while experiencing a chain of events rapidly taking place, an experience of emptiness when the baby is placed in the intensive care unit, the feeling of powerlessness when facing the real risk of the infant's death, the striking spectacle of invasive treatments, etc. The parents worry about the viability and future of their premature infant. Their parental impressions and more specifically those of the mother facing the premature birth could in and of themselves have repercussions on the development of the infant, by betting on a complex meeting and atypical interactions.

These observations have driven us to elaborate on a hypothesis that finds itself separate from the lesion model commonly applied to premature infants, and shifts the psychopathological approach to the post-traumatic reaction of the mother following the premature birth and repositions the question of behavioral disorders of the child in the interaction mother-infant field. The investigators think that the premature birth can bring about in a second phase and notably in the mother, post-traumatic symptoms as described in the post-traumatic stress state, and that this reaction could have effects on the mother-infant interactions. The investigators have carried out the current study to clarify the relationship between the mother's post-traumatic reaction triggered by the premature birth and the mother-infant interactions.

DETAILED DESCRIPTION:
2.1 Design A multicenter prospective study was performed in three French hospitals (Reims, Nancy and Besançon) between January 2008 and January 2011. The follow-up period was 18 months for each dyad.

2.2 Population

In practice, our study will be carried out in five sessions and at three visits:

The first visit in maternity service, following the birth of the child, the second visit, in the neonatology service, right before the discharge. The third time will be repeated at 6, 12 and 18 months, within the framework of the systematic tracking of premature babies within the early medico-social actions' center (CAMSP).

2.3 Data collection 2.3.1 Sociodemographic and clinical data Sociodemographic variables recorded during the study were age, marital status, level of education and profession.

For the mothers, clinical data were: number of childbirths, number of pregnancies, medical history of the pregnancy (threatened premature labor, hospitalization,...), obstetric history (miscarriage, medical interruption of pregnancy, termination of pregnancy, in vitro fertilization, threatened premature labor, prematurity, hospitalizations,…), delivery conditions (C-section or vaginal), multiple pregnancy (number of babies), anesthesia type (none, epidural, total), personal histories (medical, surgical, psychiatric, family).

For the infants, clinical data were: date of birth, term of birth, weight, size, cranial perimeter, Apgar score at five and ten minutes, necessity or not of a neonatal resuscitation, method of feeding (breast-, bottle-, mixed-feeding).

For the dyads, clinical data were the presence or absence of a specific coping (psychologist, psychomotor therapist, …).

2.3.2 Evaluation scales 2.3.2.1 For the mother Evaluation of trauma of the mother using " Perinatal Posttraumatic Stress Disorder " or PPQ.

It consists of a self--questionnaire made up of 14 items, specially adapted to the parents of perinatal high-risk children, in order to evaluate the presence of traumatic elements concerning the birth.

In order to neutralize identified biases, the investigators also evaluate the maternal co morbidity while using:

The HADS scale (Hospital Anxiety and Depression Scale) which is a self-questionnaire frequently used in international literature. Fast and easy to use, it makes it possible to evaluate anxious and depressive symptomatology of the people having somatic diseases. It makes it possible to evaluate the episodes of recent anxiety and depression and to attribute an overall score to each one. The result is expressed in a score.

The EPDS scale (Edinburgh Post-natal Depression Scale) consists of a self-questionnaire that tracks postnatal depression and includes 10 items, which the investigators offer to the mother as of the 4th week of postpartum.

The maternal social support self-evaluation by the Support Social Questionnaire (SSQ) of Sarason, proposes the measure of the number of people available and the perceived quality of this support, using 6 items.

2.3.2.2 For the child The investigators evaluate the perinatal risk of the infant with the scale Perinatal Risk Inventory (PRI). This scale uses 18 items to describe the gravity of the perinatal problems and the severity of the perinatal risk while being based on perinatal factors such as the Apgar score, the gestational age, the weight or the cranial perimeter.

The developmental evaluation of the child is done using DDST, Denver Developmental Screening Test. This assessment makes it possible to evaluate the level of the child between 0 to 6 years of age in the various fields of the development (global motricity, language, fine motricity, social contact).

The perceived temperament of the child is evaluated by the self-questionnaire filled out by the mother on the temperament of her infant QT6, translation of Bates' "Infant Characteristics Questionnaire". The mother ranks each item indicating the level of perceived difficulty in dealing with the described behavior. Four subscales have been identified through principal components analyses: Fussy/Difficult, Unadaptable, Dull, and Unpredictable.

2.3.2.3 For the interactions in the dyad Censullo's DMC (Dyadic Mutuality Code) Scale can be used for the first 6 months of the baby's life. After a 5-minute observation of the dyad interacting the observer codes 6 items (mutual attention, positive affect, reciprocity, maternal pauses, clearness of the signals of the baby, receptivity/maternal sensitivity). The score makes it possible to define a low or high interactional synchrony.

Fiese's PIPE (Pediatric Infant Parent Exam) can be used from 0 to 18 months. The mother is invited to play for a short time, games like "peek-a-boo" with her baby. The observer of the interaction grants a grade to the degree of interactional reciprocity and positive affects at the beginning, during and at the end of the play.

ELIGIBILITY:
Inclusion Criteria:

* premature birth (term ≤ to 32 weeks of amenorrhea),
* a mother with niether psychotic troubles- either acute or chronic- nor presenting an addiction (alcohol, narcotic drugs),
* a newborn with no unfavourable vital prognosis, no organic malformation and/or no genetic anomaly diagnosed,
* a mother's age ≥ 18 years,
* a native French speaker.

Exclusion Criteria:

no premature birth (term > to 32 weeks of amenorrhea),

* a mother with psychotic troubles- acute or chronic- presenting an addiction (alcohol, narcotic drugs),
* a newborn with unfavourable vital prognosis, organic malformation and/or genetic anomaly diagnosed,
* a mother's age < 18 years,
* a no native French speaker.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dyads were recruited from maternity or neonatology services.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-12-01 (Actual); Primary Completion 2010-12-01 (Actual); Study Completion 2011-08-01 (Actual)

PRIMARY OUTCOMES:
mother's post-traumatic reaction | Month 6
  relationship between the mother's post-traumatic reaction triggered by the premature birth (PPQ: Perinatal PostTraumatic Stress Disorder) and the mother-infant interactions (DMC : Dyadic Mutuality Code)

SECONDARY OUTCOMES:
relationship between the post-traumatic response of the mother in the perinatal period (PPQ: Perinatal PostTraumatic Stress Disorder) and that which is always evaluated in the mother | Month 6
relationship between perinatal risk (PRI : Perinatal Risk Inventory) and trauma (PPQ: Perinatal PostTraumatic Stress Disorder) | Month 6
relationship between pediatric assessment of the child and trauma (PPQ: Perinatal PostTraumatic Stress Disorder) | Month 6
mother's post-traumatic reaction | Month 12
  relationship between the mother's post-traumatic reaction triggered by the premature birth (PPQ: Perinatal PostTraumatic Stress Disorder) and the mother-infant interactions (PIPE : Pediatric Infant Parent Exam)
relationship between the post-traumatic response of the mother in the perinatal period (PPQ: Perinatal PostTraumatic Stress Disorder) and that which is always evaluated in the mother | Month 12
relationship between perinatal risk (PRI : Perinatal Risk Inventory) and trauma (PPQ: Perinatal PostTraumatic Stress Disorder) | Month 12
relationship between pediatric assessment of the child and trauma (PPQ: Perinatal PostTraumatic Stress Disorder) | Month 12
mother's post-traumatic reaction | Month 18
  relationship between the mother's post-traumatic reaction triggered by the premature birth (PPQ: Perinatal PostTraumatic Stress Disorder) and the mother-infant interactions (PIPE :Pediatric Infant Parent Exam)
relationship between the post-traumatic response of the mother in the perinatal period (PPQ: Perinatal PostTraumatic Stress Disorder) and that which is always evaluated in the mother | Month 18
relationship between perinatal risk (PRI : Perinatal Risk Inventory) and trauma (PPQ: Perinatal PostTraumatic Stress Disorder) | Month 18
relationship between pediatric assessment of the child and trauma (PPQ: Perinatal PostTraumatic Stress Disorder) | Month 18

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France